CLINICAL TRIAL: NCT00396786
Title: Controlled, Double-Blind, Randomized, Dose-ranging Study of Once-daily Regimen of BAY59-7939 in the Prevention of VTE in Patients Undergoing Elective Total Hip Replacement- ODIXaHIP-OD
Brief Title: Dose-ranging Study of Once-daily Regimen of BAY 59-7939 in the Prevention of VTE in Patients Undergoing Elective Total Hip Replacement
Acronym: ODIXaHIP-OD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11527; EudraCT No: 2004-001341-14
Record Dates: First submitted 2006-11-06; First posted 2006-11-07 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Venous Thromboembolism
Keywords: Prevention of venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 2 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 3 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 4 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 5 (Experimental)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 6 (Active Comparator)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Rivaroxaban 5 mg once daily plus placebo enoxaparin syringe
  Arms: Arm 1
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Rivaroxaban 10 mg once daily plus placebo enoxaparin syringe
  Arms: Arm 2
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Rivaroxaban 20 mg once daily plus placebo enoxaparin syringe
  Arms: Arm 3
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Rivaroxaban 30 mg once daily plus placebo enoxaparin syringe
  Arms: Arm 4
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Rivaroxaban 40 mg once daily plus placebo enoxaparin syringe
  Arms: Arm 5
Drug: Enoxaparin — Enoxaparin 40 mg once daily plus Rivaroxaban placebo tablets
  Arms: Arm 6

SUMMARY:
The purpose of this study is to assess different doses of a new drug (BAY 59-7939), taken as a tablet, are safe and can help prevent blood clots forming after a hip replacement operation. Patients undergoing hip replacement surgery are at risk of developing blood clots. To reduce this risk treatment to prevent clots forming is routinely given. The current treatments can include injections under the skin or other treatments that need frequent blood tests to monitor levels of drug in the body. Therefore there is a need for new drugs, which are easier to give and need less monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years or above and postmenopausal female patients
* Patients scheduled for elective primary total hip replacement (cemented or non-cemented prosthesis)
* Patients written informed consent for participation after receiving detailed written and oral previous information to any study specific procedures Exclusion Criteria:
* Related to medical history:

  * Any VTE prior to randomization
  * Myocardial infarction (MI) or TIA or ischaemic stroke within the last 6 months prior to randomisation
  * History of heparin-induced thrombocytopenia, allergy to heparins- Intracerebral or intraocular bleeding within the last 6 months prior to randomisation
* History of gastrointestinal disease with gastrointestinal bleeding within the last 6 months prior to the study
* History or presence of gastrointestinal disease which could result in an impaired absorption of the study drug (e.g. severe active inflammatory bowel disease, short gut syndrome)
* Amputation of one legRelated to current symptoms or findings:

  * Heart insufficiency NYHA class III-IV- Congenital or acquired haemorrhagic diathesis (PT INR/aPTT not within normal limits) including patients with acquired or congenital thrombopathy
  * Thrombocytopenia (platelets < 100.000/µl)- Macroscopic haematuria- Allergy to contrast media- Severe hypertension (SBP > 200 mmHg, DBP > 100 mmHg)- Impaired liver function (transaminases > 2 x ULN)
  * Impaired renal function (serum creatinine > 1.5 x ULN or creatinine clearance < 30 ml/min)
  * Active malignant disease - Presence of active peptic ulcer or gastrointestinal disease with increased risk of gastrointestinal bleeding- Body weight < 45 kg
  * Drug- or alcohol abuse- Related to current treatment- Patients who cannot stop therapy (in the opinion of the investigator/physician) with anticoagulants (e.g. phenprocoumon, warfarin-sodium, heparins and factor Xa inhibitors other than study medication) should be excluded from the study
  * Fibrinolytic therapy- Therapy with acetylic salicylic acid or other platelet aggregation inhibitors (e.g. clopidogrel, dipyridamole and ticlopidine) should be stopped one week before enrolment. Patients not able to stop ASA therapy will be excluded
  * All other drugs influencing coagulation, (exception: NSAIDs with half life < 17 hrs) will be not allowed during the study treatment period- Systemic and topical treatment with azole compounds (e.g. ketoconazole, fluconazole, itraconazole) and other strong CYP3A4-inhibitors eg HIV-protease inhibitors. Azole compounds and other strong CYP3A4-inhibitors eg HIV-protease should be stopped at least four days before enrolment
* Therapy with another investigational product within 30 days prior start of study
* Miscellaneous
* Planned intermittent pneumatic compression during active treatment period
* Planned epidural anaesthesia with indwelling epidural catheter (spinal or epidural anaesthesia without indwelling catheter are allowed)
* If traumatic or repeated epidural and spinal puncture occur the patient should be excluded from study
* Concomitant participation in another trial or study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 877 (Actual)
Dates: Start 2004-11; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Composite Endpoint of Deep Vein Thrombosis (DVT), non-fatal Pulmonary Embolism (PE) and Death from all causes | 6-10 days after surgery

SECONDARY OUTCOMES:
Incidence of DVTs (total, proximal, distal) | 6-10 days after surgery
Incidence of symptomatic Venous Thrombo Embolisms (VTEs) | 6-10 days after surgery
Incidence of major VTE (ie, Proximal DVT, PE or VTE-related death) | 6-10 days after surgery
The composite endpoint that results from the primary endpoint by substituting VTE related death for all death | 40 days
Incidence of symptomatic VTEs (total, PE, DVT) within 30 days after stop of treatment with the study drug | 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (55):
- Austria (3):
  - Wiener Neustadt, Lower Austria
  - Linz, Upper Austria
  - Vienna, Vienna
- Belgium (4):
  - Antwerp
  - Bonheiden
  - Genk
  - Hasselt
- Denmark (4):
  - Hellerup
  - Herlev
  - Hørsholm
  - Silkeborg
- France (3):
  - Paris
  - Poitiers
  - Saint-Herblain
- Germany (9):
  - Rheinfelden, Baden-Wurttemberg
  - Fürth, Bavaria
  - Garmisch-Partenkirchen, Bavaria
  - Sommerfeld, Brandenburg
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Melsungen, Hesse
  - Düsseldorf, North Rhine-Westphalia
  - Dresden, Saxony
- Israel (7):
  - Petah Tikva, Isarel
  - Haifa, Israel
  - Holon, Israel
  - Kfar Saba, Israel
  - Petah Tikva, Israel
  - Tel Aviv, Israel
  - Ẕerifin, Israel
- Italy (5):
  - Monza, Milano
  - Rozzano, Milano
  - Gubbio, Perugia
  - Bologna
  - Milan
- Netherlands (3):
  - Hilversum
  - Hoofddorp
  - Nijmegen
- Norway (3):
  - Notodden
  - Oslo
  - Rjukan
- Poland (5):
  - Bialystok
  - Gdansk
  - Krakow
  - Lublin
  - Warsaw
- Spain (4):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Valencia, Valencia
- Sweden (4):
  - Gothenburg
  - Halmstad
  - Jönköping
  - Kungälv
- London, Greater London, United Kingdom

REFERENCES:
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu